CLINICAL TRIAL: NCT05386485
Title: FUNCTION Study: Follow- Up Study iN SARS-CoV-2 infecTION. Long-term Impact on Cardiopulmonary Function and Quality of Life in Patients Recovered From SARS-CoV-2 Infection in Lima, Peru
Brief Title: Long-term Impact on Cardiopulmonary Function and Quality of Life in Patients Recovered From COVID-19.
Acronym: FUNCTION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Other Study IDs: SIDISI 203725; IN-US-983-6130 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2022-05-09; First posted 2022-05-23 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-Cov-2; Cardiovascular function; Respiratory function; Life quality; Long COVID; COVID19 Sequelae; Function test
MeSH Terms: conditions — COVID-19; Respiratory Aspiration; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 3 samples will be drawn at BL and M6 visits. Three mL of venous blood will be collected in EDTA tubes to calculate hemoglobin values using the SLS method. Four mL of venous blood will be collected in SST to calculate NT-ProBNP values using CLIA technique and the remaining serum will be stored in 1.8-ml cryovial at -70 Celsius degrees. Three mL of venous blood will be collected in EDTA tubes to separate plasma by centrifugation method and stored in 1.8-ml cryovial at -70 Celsius degrees. Plasma and serum will only be stored if it was previously authorized by the participant in the informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A (asymptomatic infection): Absence of clinical manifestation during the acute phase of SARS-CoV-2 infection until discharge.
  Interventions: Other: None intervation
- Group B1 (mild symptomatic infection): Clinical manifestation of the infection without severity signs (respiratory rate < 30/minute; peripheral oxygen saturation (SpO2) >94%) and no radiological evidence of pneumonia
  Interventions: Other: None intervation
- Group B2 (moderate symptomatic infection): Clinical manifestation of the infection without severity signs (respiratory rate < 30/minute; peripheral oxygen saturation (SpO2) >94%) and radiological evidence of pneumonia
  Interventions: Other: None intervation
- Group B3 (severe symptomatic infection): Clinical manifestation of the infection with severity signs (respiratory rate > 30/minute; peripheral oxygen saturation (SpO2) <94%) and radiological evidence of pneumonia
  Interventions: Other: None intervation
- Group B4 (critical symptomatic infection): Clinical manifestation of the infection with severity signs (respiratory rate > 30/minute; peripheral oxygen saturation (SpO2) <94%) and at least one of the following:
  I) Acute Respiratory Distress Syndrome: defined under Berlin Criteria mostly defined by a PaFi<200, II) Shock: Patient diagnosed with sepsis that despite adequate fluid resuscitation, require vasopressors to maintain a mean arterial pressure ≥65 mmHg and lactate values >2 mmol/L (>18 mg/dL) or III) Organ dysfunction that requires ICU admission
  Interventions: Other: None intervation

INTERVENTIONS:
Other: None intervation — Observational Study

SUMMARY:
FUNCTION is an observational cohort study conducted by researchers from the Instituto de Medicina Tropical Alexander von Humboldt at Universidad Peruana Cayetano Heredia and Cayetano Heredia Hospital.

The overall aim is to asses the long-term impact of SARS-CoV-2 infection on the cardiopulmonary function and quality of life in patients recovered from COVID-19, through a 6-month follow-up structured in 4 visits with clinical assessments and imaging studies performed by specialists.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following criteria (either for group A or B) in order to participate in the study:

  * Individuals of any sex over 18 years of age
  * A positive COVID-19 test result by nasopharyngeal swab for either RT-PCR or antigenic techniques within the last 14 days prior the enrollment. A laboratory-based confirmatory report will be required
  * Recruitment time close around the discharge date or no longer than 7 days after discharge
  * Group A: Individuals who had not reported signs or symptoms suggestive of COVID-19 infection
  * Group B: Individuals who had reported signs or symptoms suggestive of COVID-19 infection

Exclusion Criteria:

* An individual meeting any of the following criteria at the time of enrollment will be excluded from study participation:

  * A negative COVID-19 test result by nasopharyngeal swab for either RT-PCR or antigenic techniques
  * Known inability to keep adherent to the study (ex. incarceration, migration, travel)
  * Active pregnancy confirmed by either qualitative urine or quantitative blood beta-hCG test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients will be screened and recruited mainly from Cayetano Heredia Hospital, a tertiary-level referral center with an assigned population of nearly 3 million individuals. Also patients admitted into different public or private institutions in Lima could be considered.
  Outpatients will be screened and recruited from primary level health care centers located in different parts of Lima.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Abnormal pulmonary function | 6 months
  % of participants with carbon monoxide diffusing capacity lower than 80 percent of predicted at each study visit. The dependent variable will be categorized as dichotomic variable for subsequent analysis
Abnormal cardiovascular function | 6 months
  LVEF<50% will be considered an abnormal cardiovascular function test. The dependent variable will be categorized as dichomotoic variables for subsequent analysis.
Abnormal quality of life | 6 months
  Health-related quality of life, Medical Outcomes Study short-form (SF-36) at each visit assessed using the Short Form-36 (SF-36). The SF-36 scale consists of 8 dimensions which is subsequently converted into a percentage score. The dependent variable will be categorized as dichotomic variable for subsequent analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Cachay, MD, Principal Investigator — Universidad Peruana Cayetano Heredia; Eduardo Gotuzzo, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Instituto de Medicina Tropical Alexander von Humboldt, Universidad Peruana Cayetano Heredia, Lima Lima, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raveendran AV, Jayadevan R, Sashidharan S. Long COVID: An overview. Diabetes Metab Syndr. 2021 May-Jun;15(3):869-875. doi: 10.1016/j.dsx.2021.04.007. Epub 2021 Apr 20. PMID 33892403
- [Background] Venkataraman T, Frieman MB. The role of epidermal growth factor receptor (EGFR) signaling in SARS coronavirus-induced pulmonary fibrosis. Antiviral Res. 2017 Jul;143:142-150. doi: 10.1016/j.antiviral.2017.03.022. Epub 2017 Apr 5. PMID 28390872
- [Background] Yao XH, Li TY, He ZC, Ping YF, Liu HW, Yu SC, Mou HM, Wang LH, Zhang HR, Fu WJ, Luo T, Liu F, Guo QN, Chen C, Xiao HL, Guo HT, Lin S, Xiang DF, Shi Y, Pan GQ, Li QR, Huang X, Cui Y, Liu XZ, Tang W, Pan PF, Huang XQ, Ding YQ, Bian XW. [A pathological report of three COVID-19 cases by minimal invasive autopsies]. Zhonghua Bing Li Xue Za Zhi. 2020 May 8;49(5):411-417. doi: 10.3760/cma.j.cn112151-20200312-00193. Chinese. PMID 32172546
- [Background] Torres-Castro R, Vasconcello-Castillo L, Alsina-Restoy X, Solis-Navarro L, Burgos F, Puppo H, Vilaro J. Respiratory function in patients post-infection by COVID-19: a systematic review and meta-analysis. Pulmonology. 2021 Jul-Aug;27(4):328-337. doi: 10.1016/j.pulmoe.2020.10.013. Epub 2020 Nov 25. PMID 33262076
- [Background] Siddiqi HK, Libby P, Ridker PM. COVID-19 - A vascular disease. Trends Cardiovasc Med. 2021 Jan;31(1):1-5. doi: 10.1016/j.tcm.2020.10.005. Epub 2020 Oct 14. PMID 33068723
- [Background] Di Toro A, Bozzani A, Tavazzi G, Urtis M, Giuliani L, Pizzoccheri R, Aliberti F, Fergnani V, Arbustini E. Long COVID: long-term effects? Eur Heart J Suppl. 2021 Oct 8;23(Suppl E):E1-E5. doi: 10.1093/eurheartj/suab080. eCollection 2021 Oct. PMID 34650349
- [Background] Xie Y, Xu E, Bowe B, Al-Aly Z. Long-term cardiovascular outcomes of COVID-19. Nat Med. 2022 Mar;28(3):583-590. doi: 10.1038/s41591-022-01689-3. Epub 2022 Feb 7. PMID 35132265
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Arnold DT, Hamilton FW, Milne A, Morley AJ, Viner J, Attwood M, Noel A, Gunning S, Hatrick J, Hamilton S, Elvers KT, Hyams C, Bibby A, Moran E, Adamali HI, Dodd JW, Maskell NA, Barratt SL. Patient outcomes after hospitalisation with COVID-19 and implications for follow-up: results from a prospective UK cohort. Thorax. 2021 Apr;76(4):399-401. doi: 10.1136/thoraxjnl-2020-216086. Epub 2020 Dec 3. PMID 33273026
- [Background] Taboada M, Moreno E, Carinena A, Rey T, Pita-Romero R, Leal S, Sanduende Y, Rodriguez A, Nieto C, Vilas E, Ochoa M, Cid M, Seoane-Pillado T. Quality of life, functional status, and persistent symptoms after intensive care of COVID-19 patients. Br J Anaesth. 2021 Mar;126(3):e110-e113. doi: 10.1016/j.bja.2020.12.007. Epub 2020 Dec 10. No abstract available. PMID 33413976
- [Background] Daugherty SE, Guo Y, Heath K, Dasmarinas MC, Jubilo KG, Samranvedhya J, Lipsitch M, Cohen K. Risk of clinical sequelae after the acute phase of SARS-CoV-2 infection: retrospective cohort study. BMJ. 2021 May 19;373:n1098. doi: 10.1136/bmj.n1098. PMID 34011492
- [Derived] Cachay R, Watanabe-Tejada T, Cuno K, Gil-Zacarias M, Coombes C, Ballena I, Mejia F, Medina F, Gayoso O, Seas C, Otero L, Gotuzzo E. Long-term impact on cardiopulmonary function and quality of life among patients recovered from SARS-CoV-2 infection in a 6-month follow-up period in Lima, Peru: FUNCTION cohort study protocol. BMJ Open. 2023 Apr 20;13(4):e067365. doi: 10.1136/bmjopen-2022-067365. PMID 37080629
- See also: Pericarditis and myocarditis long after SARS-CoV-2 infection: a cross-sectional descriptive study in health-care workers. Eiros R, et al. — https://www.medrxiv.org/content/10.1101/2020.07.12.20151316v1